CLINICAL TRIAL: NCT04885829
Title: A Single Dose, Double-Blind, Two-Period, Crossover, Comparative Pharmacokinetic Study of Three Tocilizumab Products Administered by the Subcutaneous Route to Normal Healthy Volunteers
Brief Title: Comparative Study of 3 Tocilizumab Products in Normal Healthy Volunteeers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-01-002
Record Dates: First submitted 2021-05-03; First posted 2021-05-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Giant Cell Arteritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Giant Cell Arteritis | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DRL_TC (Experimental): Subcutaneous injection of DRL's Tocilizumab
  Interventions: Drug: Tocilizumab Prefilled Syringe
- RP and RMP (Active Comparator): Subcutaneous injection of Actemra and RoActemra (Commercially available Tocilizumab)
  Interventions: Drug: Tocilizumab Prefilled Syringe

INTERVENTIONS:
Drug: Tocilizumab Prefilled Syringe — 0.9ml Subcutaneous pre-filled syringes containing 162mg of Tocilizumab.
  Other Names: Actemra; RoActemra

SUMMARY:
A single dose, two period trial where participants will be given either of 3 Tocilizumab product on Day 1 during period 1 and either one of the remaining 2 Tocilizumab products on Day 1 period 2. There will be at least 6 weeks (42 days) of wash out between subsequent two period dosing. The maximum flexibility allowed between subsequent periods will be up to 9 weeks (63 days).

Names of the 3 tocilizumab products are DRL_TC, RP and RMP. So if a participant receives DRL_TC on Day 1 Period 1 then he/she will either receive RP/RMP on Day 1 Period 2.

DETAILED DESCRIPTION:
The study will be conducted at 4 sites (2 in New Zealand, 1 in Australia and 1 in India) The three pairwise product comparisons (DRL_TC vs. RP; DRL_TC vs RMP and RP vs. RMP)will be performed in parallel. Each comparison will be separately considered. Study subjectswill be randomly assigned in a 1:1:1 ratio to one of the comparisons and within eachcomparison subjects will be randomized in a 1:1 ratio to one of the two possible productsequences The total duration of the individual subject study participation will be at least 12weeks. Dosing for period 1 will be on on day 1 followed by washout out period of upto 9weeks. Dosing for Period 2 will be on Day 1.

Subjects who complete the study and are found to be positive for anti-drug antibodies (ADA)on Day 29 and/or Day 43 period 2, will be followed up every 90 days for immunogenicitysampling up to approximately one year post Period II dosing, or until two consecutive sampleshave been negative for ADA, whichever is earlier. Early dropouts will be tested forimmunogenicity at the time of EOS and if they are positive for ADAs they will be followed-up ifpossible at 90 days intervals starting from the last received dose (either Period I or Period II) ina similar manner.

300 NHV (Normal Healthy Volunteers) will be included in the study as justified under samplesize justification. After the data of these 300 volunteers become available a blinded samplesize re-estimation (BSSR) will be performed to reconfirm the statistical assumptions of thestudy design and depending upon the outcome of the BSSR, study may be stopped or thesample size may be increased, as needed to attain the required statistical power.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers, 18 to 50 years of age at the time of signing informed consent.
2. In general good health as determined by a qualified physician based on a comprehensive medical history, physical examination including vital signs, laboratory haematology, clinical chemistry, urinalysis and 12-lead ECG during screening.
3. BMI between 18.5 - 30.0 kg/m2 and body weight between 50 and 100 kg (both inclusive).
4. Screening parameters (vital signs, physical examination, clinical laboratory tests, 12-lead ECG, chest X-ray, thyroid function etc.) are within the normal range or if outside the normal range, assessed as clinically non-significant by the Investigator (unless the value constitutes an explicit exclusion criterion).
5. Male volunteers must be willing to abstain from sexual intercourse, sperm donation or willing to use in all relationships with a partner from the opposite sex a condom for the male partner and another effective method of contraception (such as an intra-uterine device, vaginal ring, oral contraceptive, injectable progesterone, or sub-dermal implant) for the female partner from the time of dosing until 3 months after the last dosing date, unless one of the partners is medically confirmed to be either infertile or surgically sterile.
6. Female volunteers should be either post-menopausal or surgically sterile. Note: ("Postmenopausal" is defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy)
7. Capable, and amenable, to provide written informed consent to the study requirements.
8. Willing to abide by study restrictions for the entire study duration.

Exclusion Criteria:

1. Positive test result for Quantiferon-TB Gold test, syphilis, hepatitis B, hepatitis C, or HIV-1 or 2.
2. Any prior exposure to tocilizumab or to any other agent directly acting on interleukin-6 or on its receptors including investigational products (e.g. siltuximab, sarilumab etc.).
3. Live virus vaccination within 3 months prior to screening or intention to receive live virus vaccination during the trial or up to 3 months after the administration of the study drug.
4. Administration of immunoglobulins for anti-tetanus and antirabies post-exposure prophylaxis within 3 weeks prior to administration of study drug.
5. History of immunodeficiency or other clinically significant immunological disorders, or auto-immune disorders, ongoing or frequent/ recurring infection defined as more than 3 per year requiring treatment or prior herpes zoster not fully healed (including the post-herpetic neuralgia period if occurring) within one year prior to randomization or history of systemic fungal infection at any time.
6. Allergy, or hypersensitivity to any recombinant human, or humanized antibodies, other therapeutic proteins, or any excipients in the study formulations.
7. Current manifestation of clinically significant (in the opinion of the Investigator) atopic allergy (e.g., asthma including childhood asthma currently showing clinical manifestations, urticaria, angioedema, eczematous dermatitis), hypersensitivity, or allergic reactions.
8. Non-suitable skin for dosing or post-dosing evaluations of upper arm (same arm to be used as the injection site in the both periods) for any reasons (including presence of tattoos, skin pigmentation disorders, scarring etc., which may obscure the injection site).
9. Blood donation, participation in any study requiring repeated blood sampling or haemorrhage requiring treatment or any transfusion in the past 3 months.
10. Screening blood pressure higher than 140 mm Hg (systolic) or higher than 90 mm Hg (diastolic) or volunteers currently on anti-hypertensive drugs. Up to two repeats on different days are allowed and, in this case, the mean of the measurements will be used to decide on eligibility. Screening blood pressure is to be measured in the sitting position after 5 minutes rest.
11. History of relevant orthostatic hypotension, fainting spells, or blackouts deemed in the opinion of the Investigator to pose clinical risk to the subjects.
12. QTc (Fridericia correction) longer than 450 milliseconds or other clinically relevant ECG abnormalities such as atrial fibrillation, atrial flutter, Wolf-Parkinson-White syndrome, or presence of a cardiac pacemaker.
13. History or presence of any clinically relevant nervous system disease including, but not restricted to any stroke/TIA (Transient Ischemic Attack), or of seizures other than febrile seizures before the age of 5 years.
14. History of and/or current gastrointestinal, renal endocrine, pulmonary, hepatic, cardiovascular (including history of or presence of angina, exertional dyspnoea, orthopnoea, congestive heart failure or myocardial infarction and thrombotic or embolic episode requiring treatment), hematological (including pancytopenia, aplastic anemia or blood dyscrasia and coagulopathies, or an INR higher than 1.5), metabolic (including known diabetes mellitus) considered as significant by the Investigator. This criterion includes any disorder or condition that, in the Investigator's opinion, may interfere with the safety of the subject, the study evaluations or the subject compliance to the study procedures and limitations.
15. ALT or AST higher than 1.25 times the ULN at screening.
16. Neutrophil count below 2 x 109/liter (2,000 per mm3) or platelet count below 100 x 109/liter (100,000 per mm3) at screening.
17. Clinically relevant hyperlipidemia (fasting serum LDL-cholesterol higher than 190 mg/dL or fasting serum triglycerides higher than 200 mg/dL or subject currently on antihyperlipidemic drugs).
18. Any active infection, even if minor, ongoing at the time of screening or dosing.
19. Presence of any non-healed wound or bone fracture of a clinically relevant size (in the Investigator's opinion).
20. Participation in an interventional or Phase I study in the last three months, or on, or participation in more than 3 studies of experimental drug products in the past 12 months, or intake of an investigational drug in another trial within 3 months or 5 half-lives (whichever is longer) prior to intake of study drug in this trial or planned intake of an investigational drug (any drug administered in a clinical trial setting is considered an investigational drug) or follow up visit scheduled from any study during the course of this trial or intake for any reason in the last 6 months of some specific long body residence drugs such as any immunoglobulin or antibody drug (except for post-exposure prophylaxis of tetanus or rabies given more than 3 weeks before the date of the first study drug dose) pirimethamine, teicoplanin, systemic retinoids, mefloquine and hydroxychloroquine.
21. History of any cancer, including carcinoma in situ, lymphoma or leukemia.
22. History of, or current intestinal ulceration or diverticulitis.
23. Major surgery within the past 12 months, major surgery planned within 12 months of study enrolment or any surgery including dental interventions planned within 3 months of study enrolment.
24. Intake of any medication including herbal products within 3 weeks prior to dosing other than for the exceptions detailed in Section 10.2-Prior and Concomitant Medications.
25. Current smokers or those who gave up smoking less than 3 months prior to screening, (thus 3 months cessation required at screening time), including alternative tobacco products such as chewing tobacco and vaping, or positive urine cotinine test at screening.
26. Positive test for alcohol in breath or drugs of abuse (including benzodiazepines, amphetamines, barbiturates, cocaine, methadone, phencyclidine 3,4-methylenedioxymethamphetamine [MDMA/ecstasy], tetrahydrocannabinol, and opiates) in urine.
27. Any history of difficulty in blood sampling or any vasovagal attack during blood sampling which in the opinion of the Investigator may relevantly interfere with the study sampling.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate the PK (Pharmacokinetics) similarity of DRL_TC vs RP, DRL_TC vs RMP and RP vs RMP. | Period I pre-dose (1hour prior to drug administration), Days 1, 2, 3, 4, 5, 6, 7, 9, 11, 15, 18, 22, 29, 36, 43 and Period II - Day 1 (dosing), 2 ,3 , 4 , 5 , 6, 7, 9, 11, 15, 18, 22, 29 , 36 , 43 (-2 to +4 days)
  AUC0-∞ and AUC0-t will be calculated
To demonstrate the PK (Pharmacokinetics) similarity of DRL_TC vs RP, DRL_TC vs RMP | Period I pre-dose (1hour prior to drug administration), Days 1, 2, 3, 4, 5, 6, 7, 9, 11, 15, 18, 22, 29, 36, 43 and Period II - Day 1 (dosing), 2 ,3 , 4 , 5 , 6, 7, 9, 11, 15, 18, 22, 29 , 36 , 43 (-2 to +4 days)
  Cmax will be calculated

SECONDARY OUTCOMES:
Safety assessment | Screening (Days -28 to -2), Day -1, predose (within 1hour before dosing), post dose (10 minutes, 60 minutes, 4 hours, 8 hours, 12 hours on day 1 and 43) and 24hours, 36hours, 48hours, 60 hours, 72 hours and 84hours after dosing
  Abnormal blood pressure
Safety assessment | Screening (Days -28 to -2), Day -1, predose (within 1hour before dosing), post dose (10 minutes, 60 minutes, 4 hours, 8 hours, 12 hours on day 1 and 43) and 24hours, 36hours, 48hours, 60 hours, 72 hours and 84hours after dosing
  Abnormal pulse rate
Safety assessment | Screening (Days -28 to -2), Day -1, predose (within 1hour before dosing), post dose (10 minutes, 60 minutes, 4 hours, 8 hours, 12 hours on day 1 and 43) and 24hours, 36hours, 48hours, 60 hours, 72 hours and 84hours after dosing
  Abnormal respiratory rate
Safety assessment | Screening (Days -28 to -2), Day -1, predose (within 1hour before dosing), post dose (10 minutes, 60 minutes, 4 hours, 8 hours, 12 hours on day 1 and 43) and 24hours, 36hours, 48hours, 60 hours, 72 hours and 84hours after dosing
  Abnormal aural temperature
Safety assessment | Screening (Day -28 to -2) to EOS visit
  Assessment of outcome of Adverse events
Safety assessment | 2,24,36,48,60,72 and 84 hours post dosing.
  Injection site reaction inspection (FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials to be used)
Safety assessment | Period I - Screening (Days -28 to -2), Day -1 (check- in), 1 (dosing),4, 5 and Period II - Day 1 (check- in), 1 (dosing) 4, 5 , 43 (-2 to +4 days)
  Normal 12 Lead ECG
Safety assessment | Period I - Screening (Days -28 to -2), check-in (day -1), 2, 5, 9, 15 and 29 and Period II - Day 1 (check- in), 2 , 5 , 9, 15, 29, 43 (-2 to +4 days)
  Abnormal Clinical laboratory data ((Total blood count including hemoglobin, hematocrit, mean corpuscular volume, leukocyte counts (total and differential), and platelet count)
Safety assessment | Period I - Screening (Days -28 to -2), check-in (day -1), 2, 5, 9, 15 and 29 and Period II - Day 1 (check- in), 2 , 5 , 9, 15, 29, 43 (-2 to +4 days)
  Abnormal Clinical lab tests (Urea, creatinine, uric acid, glucose, ALT, AST, total bilirubin (and direct if increased), sodium, potassium, chloride, calcium, total proteins, albumin, and LDH)
Safety assessment | Period I - Screening (Days -28 to -2), check-in (day -1), 2, 5, 9, 15 and 29 and Period II - Day 1 (check- in), 2 , 5 , 9, 15, 29, 43 (-2 to +4 days)
  Abnormal Clinical lab tests (Coagulation test (aPTT (Activated partial thromboplastin time) and INR (International Normalized Ratio))
Safety assessment | Period I - Screening (Days -28 to -2), check-in (day -1), 2, 5, 9, 15 and 29 and Period II - Day 1 (check- in), 2 , 5 , 9, 15, 29, 43 (-2 to +4 days)
  Abnormal Clinical lab tests (Thyroid hormones (T3, T4 and TSH))
Safety assessment | Period I - Screening (Days -28 to -2), check-in (day -1), 2, 5, 9, 15 and 29 and Period II - Day 1 (check- in), 2 , 5 , 9, 15, 29, 43 (-2 to +4 days)
  Abnormal Clinical lab tests (Lipid profile (including total, LDL and HDL Cholesterol as well as trigycerides)
Safety assessment | Period I - Screening (Days -28 to -2), check-in (day -1), 2, 5, 9, 15 and 29 and Period II - check-in (day -1), 2, 5, 9, 15, 29 ,43 (-2 to +4 days)
  Abnormal Clinical lab tests (Urine evaluation with dipstick (confirmation with microscopic examination, if abnormalities are found))
IL-6 assessment | Period I - Day-1, 2, 5, 15 and Period II - Day -1 , 2 , 5 , 15
  Change from pre-dose to selected time-points post-dose
hsCRP assessment | Period I - Day-1, 2, 5, 15 and Period II - Day -1 , 2 , 5 , 15
  Change from pre-dose to selected time-points post-dose
Neutrophil assessment | Period I - Day-1, 2, 5, 15 and Period II - Day -1 , 2 , 5 , 15
  Change from pre-dose to selected time-points post-dose
Lipid parameters assessment | Period I - Day-1, 2, 5, 15 and Period II - Day -1 , 2 , 5 , 15
  Change from baseline to selected time-points post-dose (Total, LDL, HDL and trigylcerides)
Immunogenicity assessment | Period I - On Day 1 (Randomization), 15, 29 and Period II - On day 1(Dosing)), 15, 29
  Presence of anti-drug antibodies (Confirmed positive samples, will be further tested for titre and presence of neutralizing antibodies (NAb))

CONTACTS AND LOCATIONS:
Locations (4):
- Nucleus Network, Brisbane, Brisbane, Australia
- Syngene International Ltd, Bangalore, Karnataka, India
- New Zealand (2):
  - Auckland Clinical Studies Ltd (NZCR OpCo Limited), Grafton, Auckland
  - Christchurch Clinical Studies Trust Ltd (NZCR OpCo Limited), Christchurch

IPD SHARING:
Plan to Share IPD: No